CLINICAL TRIAL: NCT03853161
Title: A Multicenter Randomized Controlled Trial Comparing High Flow Nasal Cannula and NIPPV in Preterm Infants
Brief Title: High Flow Nasal Cannula Versus Nasal Intermittent Positive Pressure (NIPPV) in Preterm Infants
Acronym: VAPORAM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Ayala Gover, principal investigator, Carmel Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMC-17-0131-CTIL
Record Dates: First submitted 2019-02-19; First posted 2019-02-25 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Preterm Infant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vapotherm arm (Experimental): Preterm infants in this arm will be given respiratory support of heated humidified high flow via Precision Flow Vapotherm, Exeter, USA
  Interventions: Other: Vapotherm
- NIPPV arm (Experimental): Preterm infants in this arm will be given respiratory support of Nasal Intermittent Positive Pressure Ventilation via the Leoni Plus neonatal ventilator
  Interventions: Other: NIPPV

INTERVENTIONS:
Other: Vapotherm — A form of non invasive ventilation used in newborns
  Other Names: Heated Humidified High Flow Nasal Cannula
  Arms: Vapotherm arm
Other: NIPPV — A form of non invasive ventilation used in newborns
  Other Names: Nasal Intermittent Positive Pressure Ventilation
  Arms: NIPPV arm

SUMMARY:
The aim of this study is to compare the effectiveness of Heated Humidified High Flow Nasal Cannula (HHHFNC) versus Nasal Intermittent Positive Pressure Ventilation (NIPPV) in preventing intubation when used as primary respiratory support for Respiratory Distress Syndrome (RDS) or post extubation in preterm infants

DETAILED DESCRIPTION:
Patient population will include preterm infants born at 24 - 36+6 weeks of gestation who are candidates for non-invasive respiratory support post extubation or as primary respiratory support after birth. They will be will be randomized to 2 groups: Heated Humidified High Flow Nasal Cannula (HHHFNC) and Nasal Intermittent Positive Pressure Ventilation (NIPPV).

This will be a prospective unblinded randomized controlled study, designed as a non-inferiority trial.

Primary outcome: The primary outcome will be rate of treatment failure (need for intubation) within 7 days of starting the study treatment

ELIGIBILITY:
Inclusion Criteria:

* Infants born at 24-27+6 weeks of gestation and up to 28 days of life who are extubated for the first time after birth or immediately after surfactant administration via (intubation-surfactant-extubation) INSURE or (minimally invasive surfactant therapy) MIST procedures.
* Infants born at 28-36+6 weeks of gestation and up to 28 days of life who are candidates for non-invasive support either as a primary modality after birth or post extubation.
* Signed parental informed consent by one of the parents

Exclusion Criteria:

* Infants who are unlikely to survive the immediate postnatal period or who have significant congenital abnormalities
* Presence of a pneumothorax prior to enrollment
* Hemodynamic instability due to sepsis or hemorrhage
* Inability to obtain parental consent
* Shortage of suitable equipment
* Infants who were intubated solely for surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2018-01-21 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Rate of intubation within 7 days of starting the study treatment | one week
  Failure of non invasive support by criteria of pH, blood carbon dioxide level, oxygen requirements or apneas

CONTACTS AND LOCATIONS:
Overall Officials: Ayala Gover, MD, Principal Investigator — Carmel Medical Center
Locations (1):
- Carmel Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No